CLINICAL TRIAL: NCT07186595
Title: A Prospective, Open-Label Study to Evaluate Subject Satisfaction With Overall Facial Appearance After Treatment With JUVÉDERM® Products in Medical Weight Loss (MWL) Subjects
Brief Title: A Study to Evaluate the Safety and Effectiveness of JUVÉDERM Products in Adult Participants for the Change of Their Overall Facial Appearance
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M25-631
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mid Face Volume Deficit
Keywords: Mid Face Volume Deficit; JUVÉDERM VOLUX XC; JUVÉDERM VOLUMA XC; JUVÉDERM VOLLURE XC; JUVÉDERM VOLBELLA XC; SKINVIVE by JUVÉDERM; JUVÉDERM ULTRA XC; JUVÉDERM ULTRA PLUS XC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open-Label JUVÉDERM (Experimental): Participants will receive at least 2 JUVÉDERM products for at least 3 indications (specific products and indications will be at the discretion of the investigator and per participant eligibility criteria) at Treatment Visit 1.
  Interventions: Device: JUVÉDERM VOLUX XC; Device: JUVÉDERM VOLUMA XC; Device: JUVÉDERM VOLBELLA XC; Device: JUVÉDERM VOLLURE XC; Device: SKINVIVE by JUVÉDERM; Device: JUVÉDERM ULTRA XC; Device: JUVÉDERM ULTRA PLUS XC

INTERVENTIONS:
Device: JUVÉDERM VOLUX XC — Injections
Device: JUVÉDERM VOLUMA XC — Injections
Device: JUVÉDERM VOLBELLA XC — Injections
Device: JUVÉDERM VOLLURE XC — Injections
Device: SKINVIVE by JUVÉDERM — Injections
Device: JUVÉDERM ULTRA XC — Injections
Device: JUVÉDERM ULTRA PLUS XC — Injections

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JUVÉDERM products in adults seeking improvement in facial volume and/or skin quality.

ELIGIBILITY:
Inclusion Criteria:

* Must meet at least 3 of the following criteria for treatment in the face with at least 2 JUVÉDERM products, per investigator's assessment:

  * Minimal, moderate, or severe on Allergan Temple Hollowing Scale (ATHS)
  * Moderate or severe for both eyes on Allergan Infraorbital Hollow Scale (AIHS)
  * Moderate or severe on Allergan Cheek Smoothness Scale (ACSS)
  * Moderate, significant, or severe on Mid-face Volume Deficit Scale (MFVDS)
  * Moderate or severe on Nasolabial Fold Severity Scale (NLFSS)
  * Minimal, mild, or moderate on Allergan Lip Fullness Scale 2 (ALFS2)
  * Moderate or severe on Allergan Chin Retrusion Scale (ACRS)
  * Moderate or severe on Allergan Loss of Jawline Definition Scale (ALJDS)
* Must be in good health as determined by subject's medical history, physical examination, and vital sign measurements.

Exclusion Criteria:

* Prior treatment with non-permanent soft tissue fillers or fat-reducing injectables in the face or neck within 12 months prior to screening.
* Excessively loose skin in the face and/or neck.
* Tendency to develop hypertrophic scarring and/or keloid scarring.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q™ Satisfaction with Facial Appearance Scale | Month 3
  The FACE-Q Satisfaction with Facial Appearance is a validated questionnaire that asks participants to report their level of satisfaction with the appearance of their face.
Number of Participants with Adverse Events (AEs) | Up to approximately Month 6
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status of Global Aesthetic Improvement on Facial Appearance Based on the Principal Investigator's Assessment Using the Global Aesthetic Improvement Scale (GAIS) | Month 3
  The GAIS uses a 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. A responder is defined as "improved" or "much improved" in the overall aesthetics assessment in the periorbital area.
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Psychological Function Scale | Month 3
  The FACE-Q Psychological Function is a validated questionnaire that asks participants to report their level of satisfaction with psychological function.
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Social Function Scale | Month 3
  The FACE-Q Social Function Scale is a validated questionnaire that asks participants to report their level of satisfaction with social function.
Change from Baseline in the Participant's Rasch-Transformed Score of the SKIN-Q Feels Scale | Month 3
  The SKIN-Q Scale is a validated questionnaire that asks participants to report their level of satisfaction with skin quality related to how the skin feels.
Change from Baseline in the Participant's Rasch-Transformed Score of the SKIN-Q Looks Scale | Month 3
  The SKIN-Q Scale is a validated questionnaire that asks participants to report their level of satisfaction with skin quality related to how the skin looks.
Percentage of Participants Achieving "Responder" Status Based on Participant Responses on the Natural Look Satisfaction Scale (NLSS) Assessment | Month 3
  The NLSS is an 8-item scale that measures satisfaction with various attributes that are associated with natural looking results following aesthetic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - Kian Aesthetic Institute /ID# 277045, Los Angeles, California
  - West Dermatology La Jolla /ID# 277034, San Diego, California
  - Pacific Clinical Innovations /ID# 277026, Vista, California
  - Skin Research Institute LLC /ID# 277038, Coral Gables, Florida
  - Monarch Plastic Surgery and Skin Renewal Center /ID# 278182, Atlanta, Georgia
  - Advanced Dermatology - Lincolnshire /ID# 277036, Lincolnshire, Illinois
  - H&H Research, LLC /ID# 277084, Metairie, Louisiana
  - DelRicht Research - New Orleans 308 /ID# 277039, New Orleans, Louisiana
  - Bellaire Dermatology Associates /ID# 278180, Bellaire, Texas
  - SkinDC /ID# 277062, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-631